CLINICAL TRIAL: NCT03184493
Title: Celebrex and Metformin for Postoperative Hepatocellular Carcinoma
Acronym: XBD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jian-Hong Zhong, Principal Investigator, Guangxi Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Celebrex for HCC
Record Dates: First submitted 2017-06-09; First posted 2017-06-12 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Celecoxib; Metformin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Celebrex (Experimental): Patients will receive celebrex (1 piece/day, 0.2mg/piece, Pfizer Pharmaceuticals Ltd) until obvious side effects.
  Interventions: Drug: Celebrex
- Metformin (Experimental): Patients will receive metformin (1 piece/bid, 250 mg/piece) until obvious side effects.
  Interventions: Drug: Metformin
- Celebrex plus Metformin (Active Comparator): Patients will receive celebrex (1 piece/day, 0.2mg/piece, Pfizer Pharmaceuticals Ltd) until obvious side effects. In addition, patients will receive metformin (1 piece/bid, 250 mg/piece) until obvious side effects.
  Interventions: Drug: Celebrex plus Metformin
- Empty control group (No Intervention): This group patients will not receive any postoperative adjuvant therapy.

INTERVENTIONS:
Drug: Celebrex plus Metformin — This group patients will receive metformin and celebrex.
  Arms: Celebrex plus Metformin
Drug: Celebrex — This group patients will receive celebrex.
  Arms: Celebrex
Drug: Metformin — This group patients will receive metformin.
  Arms: Metformin

SUMMARY:
This prospective trial aims to compare the role of celebrex alone, metformin alone, and celebrex plus metformin in preventing HCC recurrence after hepatic resection.

DETAILED DESCRIPTION:
Hepatic resection is a popular curative treatment for patients with early-stage HCC and well-preserved liver function. Although overall survival after resection has been increasing, the median 5-year disease-free survival rate after resection remains at only about 37% for early-stage HCC. In fact, the 5-year recurrence rate is as high as 74% for intermediate and advanced HCC. Postoperative recurrence may be due to intrahepatic metastasis arising from the primary tumor or it may be de novo metastasis (multicentric) that arises spontaneously in the residual liver. Intrahepatic metastasis is the primary mechanism of early recurrence, which occurs <2 years after resection; multicentric metastasis is the principal mechanism behind late recurrence, which occurs at least 2 years after resection.

In the past few years, some observational studies with small sample size found metformin and celebrex (selective cyclic oxidase-2 inhibitors) may reduce the rate of HCC after surgery. However, no prospective study compare their efficacy in preventing HCC recurrence. This trial aims to compare the role of celebrex alone, metformin alone, and celebrex plus metformin in preventing HCC recurrence after hepatic resection.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Diagnosis of HCC was confirmed by histopathological examination of surgical samples in all patients
* Patients have Child-Pugh A or B liver function
* No previous neoadjuvant treatment
* No evidence of macrovascular invasion, metastasis to the lymph nodes and/or distant metastases on the basis of preoperative imaging results and perioperative findings
* No malignancy other than HCC for 5 years prior to the initial HCC treatment

Exclusion Criteria:

* History of cardiac disease
* Known history of human immunodeficiency virus (HIV) infection
* Known Central Nervous System tumors including metastatic brain disease
* History of organ allograft
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study Pregnant or breast-feeding patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-06-02 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with tumor recurrence | 1-year
  The 1-year tumor recurrence will be compared between the three groups

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Tumor Hospital of Guangxi Medical University, Nanjing, Guangxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhong JH, Ma L, Li LQ. Postoperative therapy options for hepatocellular carcinoma. Scand J Gastroenterol. 2014 Jun;49(6):649-61. doi: 10.3109/00365521.2014.905626. Epub 2014 Apr 10. PMID 24716523
- [Background] Ling S, Song L, Fan N, Feng T, Liu L, Yang X, Wang M, Li Y, Tian Y, Zhao F, Liu Y, Huang Q, Hou Z, Xu F, Shi L, Li Y. Combination of metformin and sorafenib suppresses proliferation and induces autophagy of hepatocellular carcinoma via targeting the mTOR pathway. Int J Oncol. 2017 Jan;50(1):297-309. doi: 10.3892/ijo.2016.3799. Epub 2016 Dec 9. PMID 27959383
- [Background] Kim G, Jang SY, Han E, Lee YH, Park SY, Nam CM, Kang ES. Effect of statin on hepatocellular carcinoma in patients with type 2 diabetes: A nationwide nested case-control study. Int J Cancer. 2017 Feb 15;140(4):798-806. doi: 10.1002/ijc.30506. Epub 2016 Nov 16. PMID 27861855
- [Background] Chan KM, Kuo CF, Hsu JT, Chiou MJ, Wang YC, Wu TH, Lee CF, Wu TJ, Chou HS, Lee WC. Metformin confers risk reduction for developing hepatocellular carcinoma recurrence after liver resection. Liver Int. 2017 Mar;37(3):434-441. doi: 10.1111/liv.13280. Epub 2016 Nov 13. PMID 27775209
- [Background] Zhou YY, Zhu GQ, Liu T, Zheng JN, Cheng Z, Zou TT, Braddock M, Fu SW, Zheng MH. Systematic Review with Network Meta-Analysis: Antidiabetic Medication and Risk of Hepatocellular Carcinoma. Sci Rep. 2016 Sep 19;6:33743. doi: 10.1038/srep33743. PMID 27642100
- [Background] Tong H, Wei B, Chen S, Xie YM, Zhang MG, Zhang LH, Huang ZY, Tang CW. Adjuvant celecoxib and lanreotide following transarterial chemoembolisation for unresectable hepatocellular carcinoma: a randomized pilot study. Oncotarget. 2017 Jul 18;8(29):48303-48312. doi: 10.18632/oncotarget.15684. PMID 28430638
- [Background] Tong H, Li X, Wei B, Tang C. Combinative treatment of transarterial chemoembolization, celecoxib and lanreotide in unresectable hepatocellular carcinoma. Clin Res Hepatol Gastroenterol. 2015 Oct;39(5):e65-6. doi: 10.1016/j.clinre.2015.01.008. Epub 2015 Mar 4. No abstract available. PMID 25746137